CLINICAL TRIAL: NCT04581512
Title: A Modular, Multipart, Multi-arm, Open-label, Phase I/IIa Study to Evaluate the Safety and Tolerability of EP0042 Alone and in Combination With Anti-cancer Treatments in Patients With Advanced Malignancies
Brief Title: Study to Evaluate the Safety and Tolerability of EP0042
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ellipses Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP0042-101
Record Dates: First submitted 2020-09-16; First posted 2020-10-09 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes | interventions — venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Module 1 EP0042 (Experimental): Establishing the safety of EP0042 as a monotherapy and establishing an appropriate dose to take forward into subsequent modules.
  Interventions: Drug: EP0042
- Module 2 EP0042 (Experimental): * Part A: To evaluate the safety, tolerability, of EP0042 + a Bcl-2 inhibitor (venetoclax) in patients with R/R FLT3 wildtype (WT) AML.
  * Part B: To evaluate the safety, tolerability, of EP0042 in combination with a Bcl 2 inhibitor (venetoclax) + a hypomethylating agent (azacitidine) in patients with R/R FLT3 WT or newly diagnosed AML.
  Interventions: Drug: EP0042; Drug: Venetoclax; Drug: Azacitidine (AZA)

INTERVENTIONS:
Drug: EP0042 — EP0042 Oral 20 mg 50 mg capsules
Drug: Venetoclax — Venetoclax
  Arms: Module 2 EP0042
Drug: Azacitidine (AZA) — Azacitidine
  Arms: Module 2 EP0042

SUMMARY:
A research study looking at a new treatment for patients with advanced cancer, to investigate different doses of the experimental study drug, EP0042, in order to determine a dose, which is safe, well-tolerated and likely to be effective in treating AML (acute myeloid leukaemia).

ELIGIBILITY:
General

1. Male or female patients aged ≥ 18 years of age, at the time of informed consent, with histological or cytological confirmation of AML
2. Ability to understand and provide written informed consent before any study-specific procedures, sampling, or analyses, including access to archival tumor tissue
3. Ability to swallow and retain oral medication
4. Sufficient life expectancy to allow the patient to complete at least 1 cycle (28 days) of the treatment period.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2 at screening
6. In the opinion of the investigator, all other relevant medical conditions must be well-managed and stable for at least 28 days prior to first administration of study drug
7. Patients with pathologically confirmed/documented AML or MDS, as defined by the 2022 European LeukaemiaNet (ELN) recommendations, or CMML, as defined by World Health Organization (WHO) criteria, who have relapsed from or are refractory to previous therapy and have failed all (or are not eligible for/intolerant to) available approved therapies for their disease.
8. Patients with relapsed/refractory FLT3 WT AML.
9. Previous exposure to venetoclax, hypomethylating agent and/or FLT3 inhibitors (gilteritinib, midostorin, quizartinib, sorafenib) is allowed for relapsed/refractory AML patients.
10. Mutation status of patients must be known at trial entry.
11. Female patients should either be of non-child-bearing potential or must agree to use highly effective methods of contraception from Screening until 6 months following administration of the last dose of study drug
12. Male patients must use double barrier contraception from enrolment through treatment and for 6 months following administration of the last dose of study drug

5.2 Core Exclusion Criteria

Patients with any of the following will not be included in the study:

Disease Under Study and Prior Anticancer Treatment

1. Suspected brain and/or leptomeningeal metastases that are symptomatic or untreated or that require current therapy
2. Acute promyelocytic leukemia (FAB:M3)
3. Systemic anti-cancer therapy for the disease under study within 2 weeks of the first dose of study treatment. If the previous anti-cancer therapy has a very long half-life and may interact with EP0042, e.g. a strong CYP3A4 inhibitor, the washout period may need to be increased for safety reasons but will be no longer than 3 weeks (Concomitant hydroxyurea is acceptable and will be permitted throughout the screening period and during first 6 cycles of study treatment)
4. Ongoing toxic manifestations of previous treatments that have not reduced to at least CTCAE Grade 1. Exceptions to this are alopecia or certain Grade 2 treatment related toxicities, which in the opinion of the Investigator should not exclude the patient.
5. Transplantation (allogeneic or autologous) within last 90 days, or on active immunosuppressive therapy for graft versus host disease in last 2 weeks

   Laboratory Parameters
6. Patient with any out-of-range laboratory values defined as shown below.

   • Creatinine clearance (calculated using Cockcroft-Gault formula, or measured) < 50 mL/ min
7. Inadequate liver function as demonstrated by

   * total serum bilirubin ≥ 1.5 times the upper limits of normal range (ULN) or
   * ALT ≥3 times the ULN or
   * AST ≥3 times the ULN or
   * AST or ALT ≥5 times the ULN in the presence of liver involvement by leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) from the first dose through the end of the DLT observation period. | First cycle of treatment (28 Days)
  Incidence of dose-limiting toxicities (DLT)

CONTACTS AND LOCATIONS:
Overall Officials: David Taussig, Principal Investigator — The Royal Marsden, UK
Locations (6):
- Royal Perth Hospital, Perth, Western Australia, Australia
- Netherlands (2):
  - Amsterdam UMC, Amsterdam, Amsterdam
  - Erasmus MC, Rotterdam, Rotterdam
- United Kingdom (3):
  - University College London Hospital, London, London
  - The Royal Marsden, London, UK
  - The Christie Hospital, Manchester

IPD SHARING:
Plan to Share IPD: No